CLINICAL TRIAL: NCT05721963
Title: Clinical Study on the Accuracy of Proteomics in Evaluating Lymph Node Metastasis Status and Comparation With Pathological Examination in Cholangiocarcinoma Patients
Brief Title: Study on the Accuracy of Proteomics in Evaluating Lymph Node Metastasis Status in Cholangiocarcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-087-01
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Lymph Node Metastasis; Proteomics
MeSH Terms: conditions — Cholangiocarcinoma; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Resected lymph node samples will be profiled by proteomic approaches for lymph node metastasis status evaluation. And the residual samples will be kept in liquid nitrogen for a specific time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University: The cohort of Sun Yat-Sen Memorial Hospital of Sun Yat-sen University is the exploration cohort.
  Interventions: Diagnostic Test: No interventions.

INTERVENTIONS:
Diagnostic Test: No interventions. — No interventions.

SUMMARY:
This is a single-center, prospective, observational and exploratory clinical study. The object of this study is to evaluate the accuracy of proteomics approaches on resected lymph node samples in evaluating lymph node metastasis status in cholangiocarcinoma patients.

DETAILED DESCRIPTION:
The current gold standard for the diagnosis of lymph node metastasis is pathological examination of surgically resected lymph node specimens. However, lymph node metastases are different from the primary lesions, and the distribution of tumor cells is heterogeneous and more dispersed. Therefore, a single thin pathological section is difficult to obtain complete information, which may be misdiagnosed due to the failure to examine on the section containing tumor cells or the presence of micro-metastases.

The application of proteomics can obtain the overall information of the samples, including the remodeling of the microenvironment by the tumor metastases and the acclimation even before the metastasis, resulting in significant changes in the protein expression profiles of the lymph nodes, which are difficult to be completely presented in conventional pathological sections. This study aims to evaluate the accuracy of proteomics approaches on resected lymph node samples in evaluating lymph node metastasis status in cholangiocarcinoma patients, assisting in guiding precision medicine and making therapeutic decisions.

Positive controls of lymph node metastases and negative controls of normal lymph nodes were previously profiled using proteomic approaches. Machine-learning clustering method will be used to classify the newly examined lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* The patient must sign an informed consent form;
* Age 18-75 years old, both male and female;
* ECOG performance status score (PS score) 0-2;
* Child-Pugh score A period;
* Have not received any systemic treatment within 6 months;
* The functional indicators of important organs meet the following requirements (1)Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; (2)Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range; (3)Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; (4)Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula);
* For women who are not breastfeeding or pregnant, use contraception during treatment or 12 months after the end of treatment.

Exclusion Criteria:

* Unresectable cholangiocarcinoma patients or postoperative diagnosis of cholangiocarcinoma recurrence and metastasis;
* Past or simultaneous suffering from other malignant tumors;
* Have used gemcitabine-based chemotherapy or radiotherapy within 6 months;
* Severe cardiopulmonary and renal dysfunction;
* Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements);
* Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
* After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000;
* A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
* Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period;
* Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
* A history of psychotropic drug abuse, alcohol or drug abuse;
* Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed cholangiocarcinoma patients who underwent radical resection and lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis status of each examined lymph nodes by pathological tests | 1 month
  The pathological examination results of each resected lymph nodes will be recorded
Lymph node metastasis status of each lymph nodes evaluated by proteomic approaches | 2 month
  Machine-learning clustering will be applied to classify the lymph node metastasis status of each lymph nodes based on proteomic profiles

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No